CLINICAL TRIAL: NCT00948363
Title: The Effect of Kiwi on Blood Pressure, Endothelial Function, Antioxidant Capacity and Gene Expression in Mildly Hypertensive Subjects
Brief Title: The Effect of Kiwi on Blood Pressure, Endothelial Function, Antioxidant Capacity and Gene Expression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Tor Ole Klemsdal, Chief Consultant, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1335
Record Dates: First submitted 2009-07-27; First posted 2009-07-29 (Estimated); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Hypertension
Keywords: Kiwi fruits; Blood pressure; Endothelial function; Antioxidant capacity
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Kiwi fruits (Active Comparator)
  Interventions: Other: Kiwi fruits
- Apple (Placebo Comparator)
  Interventions: Other: Apple

INTERVENTIONS:
Other: Kiwi fruits — Daily intake of 3 kiwi fruits for 8 weeks
  Arms: Kiwi fruits
Other: Apple — Daily intake of 1 apple (equivalent in energy) for 8 weeks
  Arms: Apple

SUMMARY:
The purpose of this study is to determine whether the intake of kiwi fruits will reduce systolic and diastolic blood pressure compared to intake of apples. The investigators hypothesize that the increased intake lutein or other components in the kiwi fruit will enhance nitric oxide bioavailability and lead to vascular relaxation.

DETAILED DESCRIPTION:
An interesting finding in the Oslo Antioxidant Study was that intake of 3 kiwi fruits reduced blood pressure in a clinical significant manner compared to controls. The mechanism for the blood pressure reducing effect of kiwi or the responsible components are not elucidated. However, plasma lutein levels and antioxidant capacity measured by the ferric reducing antioxidant power was increased in the kiwi group. Moreover, gene expression was also altered by the increased intake of kiwi.

ELIGIBILITY:
Inclusion Criteria:

* Systolic blood pressure 130-159 mmHg
* Diastolic blood pressure 85-99 mmHg
* Body mass index <35 kg/m2

Exclusion Criteria:

* Systolic blood pressure >160 mmHg or <129 mmHg
* Diastolic blood pressure >100 mmHg or <84 mmHg
* Current use or need for blood pressure lowering medication
* Symptomatic cardiovascular disease, diabetes, renal dysfunction, psychiatric disorder, pregnancy or lactation, history of obesity surgery.

Ages: 35 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2009-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 8 weeks

SECONDARY OUTCOMES:
Endothelial function | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Serena Tonstad, Professor, Principal Investigator — Preventive Cardiology, Oslo University Hospital
Locations (2):
- Norway (2):
  - Department of Preventive Cardiology, Oslo
  - Oslo University Hospital, Oslo

REFERENCES:
- [Derived] Svendsen M, Tonstad S, Heggen E, Pedersen TR, Seljeflot I, Bohn SK, Bastani NE, Blomhoff R, Holme IM, Klemsdal TO. The effect of kiwifruit consumption on blood pressure in subjects with moderately elevated blood pressure: a randomized, controlled study. Blood Press. 2015 Feb;24(1):48-54. doi: 10.3109/08037051.2014.976979. Epub 2014 Dec 8. PMID 25483553